CLINICAL TRIAL: NCT04054778
Title: A Randomized Controlled Trial Comparing Avatar Therapy to Cognitive Behavioral Therapy in Schizophrenia With Treatment Refractory Hallucinations
Brief Title: Comparaison of Avatar Therapy to Cognitive Behavioral Therapy in Schizophrenia With Treatment Refractory Hallucinations
Acronym: Phase3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Alexandre Dumais, Psychiatrist, Clinical Associate Professor, Principal Investigator, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-12-2019-1726
Record Dates: First submitted 2019-06-19; First posted 2019-08-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Auditory Hallucination, Verbal; Treatment-resistant Schizophrenia
Keywords: Auditory verbal hallucinations; Schizophrenia; Treatment-resistant; Psychotherapy; Cognitive Behavioral Therapy; Avatar Therapy; Virtual reality
MeSH Terms: conditions — Hallucinations; Schizophrenia, Treatment-Resistant; Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized to receive either TA or CBTp.
Who Masked: Outcomes Assessor
Masking Description: The therapists, the study coordinator and the participants will be aware of the interventions after the allocation randomization. The principal investigators and independent evaluators will be blind to the random allocation conditions. The evaluators will be separated from the therapists by working at a separate location on the hospital grounds and will sign agreements not to discuss cases with any other team member. Management of the evaluations will be delegated to a coordinator preventing any direct contact between the investigators and the independent evaluators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatar Therapy (Experimental): Participants will be offered 9 individual and weekly sessions of 1 hour, which will be administered in an individual format by a licensed psychologist or psychiatrist experienced with psychosis patients. The therapy will consist in prompting participants to enter in a dialogue with their persecutor to better regulate their emotional responses. Over the course of the therapy, the avatar's speech and tone will gradually be changed by the therapist to echo participants' improved ability to regulate their emotions. That is, the avatar will progressively change from being abusive to becoming helpful and supportive. By doing so, the therapy will seek to reinforce participants' feeling of empowerment over their voices.
  Interventions: Behavioral: Avatar Therapy
- Cognitive Behavioral Therapy (Active Comparator): Participants will be offered 9 individual and weekly sessions of 1 hour, which will be administered in an individual format by a licensed psychologist or psychiatrist trained in Cognitive Behavioral Therapy for psychosis (CBTp). The program is derived and adapted from current evidence-based treatments for hallucinations. The 9 CBTp sessions will consist of a succession of learning modules and suggested task assignments.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Avatar Therapy — Participants will be offered 9 individual and weekly sessions of 1 hour, which will be administered in an individual format by a licensed psychologist or psychiatrist experienced with psychosis patients. The therapy will consist in prompting participants to enter in a dialogue with their persecutor to better regulate their emotional responses. Over the course of the therapy, the avatar's speech and tone will gradually be changed by the therapist to echo participants' improved ability to regulate their emotions. That is, the avatar will progressively change from being abusive to becoming helpful and supportive. By doing so, the therapy will seek to reinforce participants' feeling of empowerment over their voices.
  Arms: Avatar Therapy
Behavioral: Cognitive Behavioral Therapy — Participants will be offered 9 individual and weekly sessions of 1 hour, which will be administered in an individual format by a licensed psychologist or psychiatrist trained in Cognitive Behavioral Therapy for psychosis (CBTp). The program is derived and adapted from current evidence-based treatments for hallucinations. The 9 CBTp sessions will consist of a succession of learning modules and suggested task assignments.
  Other Names: CBT for psychosis
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Schizophrenia is associated with long-lasting health, social and financial burden for patients, families, caregivers and society. According to the World Health Organization, this burdensome illness is one of the top 10 causes of disability in developed countries. The costs associated with hospitalization, lifelong treatment and loss of productivity lead to a great economic burden. In Canada, the total annual costs associated with schizophrenia are over $10 billion. The main reason for this heavy burden is that 25-30% of schizophrenia patients respond very poorly to antipsychotic medication. Moreover, psychotherapeutic treatment alternatives are very limited for this suffering population. This unmet clinical need requires innovation and action. Psychotherapeutic treatment alternatives such as Cognitive Behavior Therapy (CBT) are very limited and provide at best moderate results. Virtual reality (VR) opens new exciting avenues to treat this illness. With immersive VR, our team recently tested a novel psychotherapeutic intervention, Avatar Therapy (AT), where the therapist engages in a dialogue with the patient through a virtual representation of their distressing voice. This relational and experiential approach offers a unique opportunity to help patients gain control over their voice. The preliminary results of our randomized-controlled trial (RCT) pilot showed a large effect on auditory verbal hallucination for AT and a moderate effect for CBT. The main goal of the currently proposed RCT study will be to examine if AT is superior to CBT for the treatment of chronic auditory hallucinations in schizophrenia. As evidence-based therapeutic options are limited for this burdensome illness and provide only modest symptomatic relief, the current trial will contribute to the validation of a novel approach answering a fundamental clinical need. The demonstration of the superior efficacy of AT would be a great breakthrough and will open new avenues to clinical treatment.

DETAILED DESCRIPTION:
Schizophrenia is associated with long-lasting health, social and financial burden for patients, families, caregivers and society. According to the World Health Organization, this burdensome illness is one of the top 10 causes of disability in developed countries. The costs associated with hospitalization, lifelong treatment and loss of productivity lead to a great economic burden. In Canada, the total annual costs associated with schizophrenia are over $10 billion. The main reason for this heavy burden is that 25-30% of schizophrenia patients respond very poorly to antipsychotic medication. Moreover, psychotherapeutic treatment alternatives are very limited for this suffering population. This unmet clinical need requires innovation and action. Psychotherapeutic treatment alternatives such as Cognitive Behavior Therapy (CBT) provide at best moderate results. Using immersive virtual reality, our team recently tested a novel psychotherapeutic intervention, Avatar Therapy (AT), where the therapist engages in a dialogue with the patient through a virtual representation of the patient's distressing voice. This approach, being both relational and experiential, provides a unique opportunity to aid patients gain control over their voice. The results of our pilot study on AT were clinically promising for the severity and distress related to hallucinations, positive symptomatology and emotion regulation. The preliminary results of our small pilot randomized-controlled trial showed a large effect of AT on auditory verbal hallucination, while a moderate effect was found for our adapted short CBT for hallucinations. To further research in this field, the primary goal of this single-blinded randomized-controlled, single-site parallel study is to show that AT is superior to CBT for the treatment of persistent auditory hallucinations in schizophrenia. The secondary goal is to examine the effects of these interventions on emotion regulation, mood symptoms (anxiety and depression), self-esteem, level of functioning and quality of life. To do so, each treatment group will include 68 participants over 18 years of age hearing persecutory voices and suffering from treatment resistant schizophrenia or schizoaffective disorder. AT comprises of 9 weekly sessions: 1 avatar creation session and 8 therapeutic sessions, where the patients are confronted to their reproduced hallucinatory experience and are encouraged to enter in a dialogue with their virtual persecutor. CBT includes 9 weekly sessions consisting of learning modules and task assignments. Subjects will be evaluated at pre- and post-treatment. Follow-ups will be ensured at 3, 6 and 12 months to assess primary (auditory hallucination) and secondary outcomes. Mixed model analyses will be performed to measure and compare the effects of both interventions. As evidence-based therapeutic options are limited for this burdensome illness and provide only modest symptomatic relief, the current trial will contribute to the validation of a novel approach answering a fundamental clinical need. Ultimately, the demonstration of the superior efficacy of AT would be a great breakthrough and will open new avenues to clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of schizophrenia or schizoaffective disorder
* Distressing auditory verbal hallucinations
* Did not respond to 2 antipsychotic trials
* Stable doses of medication during the last 2 months prior to enrollment

Exclusion Criteria:

* Substance use disorder within the last 12 months
* Neurological disorder
* Intellectual disability
* Unstable and serious physical illnesses
* Experiencing an acute psychotic episode
* Cognitive Behavioral Therapy for psychosis within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Psychotic Symptom Rating Scale - Auditory Hallucinations | Within 1 week after treatment (compared with 1 week before treatment)
  Psychotic Symptom Rating Scale - Auditory Hallucinations: 11-item structured interview assessing the severity of auditory hallucinations (scale 0-44); Subscales: Frequency (0-12), Distress (0-20); higher values = worse

SECONDARY OUTCOMES:
Change in the Beliefs About Voices Questionnaire - Revised | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Beliefs About Voices Questionnaire - Revised: 35-item self-report measure designed to assess key beliefs and responses people have concerning their voice (0-105); Subscales: Malevolence (0-18), Omnipotence (0-18), Benevolence (0-18); higher scores = worse
Change in the Positive And Negative Syndrome Scale | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Positive And Negative Syndrome Scale: 30-item semi-structured interview investigating overall symptoms severity of schizophrenia in the last week; Subscales: Positive (7-49), Negative (7-49), General (16-112), Total score (subscales summed; 30-210); higher values = worse symptomatology
Change in the Calgary Depression Scale for schizophrenia | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Calgary Depression Scale for schizophrenia: 9-item semi-structured scale to assess the level of depression in schizophrenia (total score range: 0-27; higher values = worse depressive symptoms)
Change in the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form: 16-item self-report scale measuring enjoyment and satisfaction experienced during the past week in various areas of daily functioning (16-80); higher values = better
Change in the Quality of life scale | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  Quality of life scale: 21-item semi-structured scale measuring quality of life (0-126); higher score = better quality of life
Change in Igroup Presence Questionnaire | During the therapy (at the end of the first and last session of Avatar Therapy)
  Igroup Presence Questionnaire: 14-item scale measuring the sense of presence; higher score = better presence
Change in the Psychotic Symptom Rating Scale - Auditory Hallucinations | Follow-ups at 3 months, 6 months and 12 months (compared with 1 week before treatment and with 1 week after treatment))
  Psychotic Symptom Rating Scale - Auditory Hallucinations: 11-item structured interview assessing the severity of auditory hallucinations; Subscales: Frequency (0-12), Distress (0-20); higher score = worse

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Dumais, MD, PhD, Principal Investigator — Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Locations (1):
- Centre de recherche de l'Institut universitaire en santé mentale de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT04054778/Prot_SAP_001.pdf